CLINICAL TRIAL: NCT06752525
Title: Opioid Sparing Effect of Sphenopalatine Ganglion Block in Functional Endoscopic Sinus Surgery: a Randomized Controlled Clinical Trial.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ali Ismaeil, resident doctor at Assiut University hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPGB sinus surgery
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Sinus Surgery
Keywords: sphenopalatine ganglion block
MeSH Terms: interventions — Bupivacaine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): patients will receive SPGB block with 2 ml volume on each side (1.5 mL of bupivacaine 0.5% + 0.5 mL of magnesium sulphate 10%)
  Interventions: Drug: Bupivacaine; Drug: Magnesium Sulphate 500 mg
- group B (Experimental): patients will receive SPGB block with 2 ml volume on each side (1.5 ml bupivacaine 0.5% plus 0.5 ml saline).
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — patients will receive SPGB block with 2 ml volume on each side (1.5 mL of bupivacaine 0.5% + 0.5 mL of magnesium sulphate 10%).
Drug: Magnesium Sulphate 500 mg — patients will receive SPGB block with 2 ml volume on each side (1.5 ml bupivacaine 0.5% plus 0.5 ml saline).
  Arms: Group A

SUMMARY:
Functional endoscopic sinus surgery (FESS) is widely recognized as a safe and preferred treatment option for various conditions, particularly nasal polyps and rhinosinusitis . This technique has been shown to improve postoperative symptoms by 86.3% in patients with chronic inflammatory paranasal sinus diseases .

The aim of this study is to evaluate the effect of adding of MgSO4 to bupivacaine via SPGB block for postoperative pain for 24 hours in patients scheduled for FESS as opioid free anaesthesia.

DETAILED DESCRIPTION:
However, managing postoperative pain remains a significant challenge. Research suggests that 86% of surgical patients experience pain, with 75% enduring moderate to severe levels .

The Sphenopalatine Ganglion Block (SPGB) is an effective, safe, and well-tolerated method for managing craniofacial pain. The ganglion comprises both sensory and autonomic nerves, which innervate the nasal cavity, palate, and certain areas of the nasopharynx and oropharynx . SPGB involves the administration of analgesic agents into the nasal cavity, typically through an endoscopic approach due to the challenges of transnasal injection . Some complications, such as postoperative nosebleeds, and temporary numbness of the palate, have been observed following the blockade with endoscopic intervention, but these are generally temporary .

Studies evaluating the effects of the sphenopalatine block in endoscopic sinus surgery suggest that patients who received the ganglion block experienced reduced postoperative pain compared to those in the placebo group when combined with general anaesthesia .

ELIGIBILITY:
Inclusion Criteria:

* • Patients programmed for elective FESS

  * American society of anaesthesiologists (ASA) physical state I-II
  * Age over 18 years and less than 60-years-old.

Exclusion Criteria:

* • Known hypersensitivity to the study drugs.

  * Inability to accurately describe postoperative pain to investigators.
  * Opioid tolerance or dependence.
  * Patient refusal
  * History of renal, liver, cardiac, neuropsychiatric disorder problems.
  * Bleeding or coagulation abnormality.
  * Infection at the site of injection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain according to (NRS) | 24 hours
  The effect of adding of MgSO4 to bupivacaine via SPGB block for postoperative pain according to (NRS) for 24 hours in patients scheduled for FESS

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Qudah M. Endoscopic sphenopalatine ganglion blockade efficacy in pain control after endoscopic sinus surgery. Int Forum Allergy Rhinol. 2016 Mar;6(3):334-8. doi: 10.1002/alr.21644. Epub 2015 Sep 15. PMID 26370724
- [Background] Kesimci E, Ozturk L, Bercin S, Kiris M, Eldem A, Kanbak O. Role of sphenopalatine ganglion block for postoperative analgesia after functional endoscopic sinus surgery. Eur Arch Otorhinolaryngol. 2012 Jan;269(1):165-9. doi: 10.1007/s00405-011-1702-z. Epub 2011 Jul 8. PMID 21739090
- [Background] Cho DY, Drover DR, Nekhendzy V, Butwick AJ, Collins J, Hwang PH. The effectiveness of preemptive sphenopalatine ganglion block on postoperative pain and functional outcomes after functional endoscopic sinus surgery. Int Forum Allergy Rhinol. 2011 May-Jun;1(3):212-8. doi: 10.1002/alr.20040. Epub 2011 Apr 13. PMID 22287376
- [Background] Sanders M, Zuurmond WW. Efficacy of sphenopalatine ganglion blockade in 66 patients suffering from cluster headache: a 12- to 70-month follow-up evaluation. J Neurosurg. 1997 Dec;87(6):876-80. doi: 10.3171/jns.1997.87.6.0876. PMID 9384398
- [Background] Xiong BJ, Xu Y, Jin GL, Liu M, Yang J, Yu CX. Analgesic effects and pharmacologic mechanisms of the Gelsemium alkaloid koumine on a rat model of postoperative pain. Sci Rep. 2017 Oct 27;7(1):14269. doi: 10.1038/s41598-017-14714-0. PMID 29079733
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004